CLINICAL TRIAL: NCT01761123
Title: An Open Label Phase I Substudy to Evaluate the Safety and Ability to Enhance Immunogenicity of VXA-A1.1 by Delivery Directly to the Ileum Using the InteliSite Companion Capsule in Healthy Adult Males
Brief Title: Immunogenicity of Seasonal Influenza by Delivery Directly to Ileum
Acronym: ICC H1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VXA02-002
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Seasonal Influenza
Keywords: Prevention of Influenza

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VXA-A1.1 (Experimental): Intestinal Delivery
  Interventions: Biological: VXA-A1.1

INTERVENTIONS:
Biological: VXA-A1.1

SUMMARY:
the purpose of the study is to determine the safety and tolerability of VXA-A1.1, an adjuvanted adenoviral based influenza vaccine, when delivery is targeted to the ileum, using a radio controlled capsule. The secondary objective is to evaluate the immune response (cellular and humoral) of two doses of VXA-A1.1 oral vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete informed consent
* Healthy, as established by medical history, physical exam, and laboratory assessments
* Has normal bowel movements
* Willing to abstain from caffeine and xanthine containing substances for 24 hours before procedure until after discharge

Exclusion Criteria:

* Not able to donate up to 550 ml of blood over several months
* Exposure to an investigational drug or vaccine 8 weeks prior to study
* Abnormal ECG findings
* History of irritable bowl or any other inflammatory gastrointestinal disorder
* Any individual with increased risk for bowl obstruction
* Radiation exposure above target values 50 mSv within the past 30 days or a cumulative dose above 150 mSV in the past 12 months
* History of substance abuse
* Subject unwilling to use an approved method of contraception during study and for 2 months after study
* Positive for HCV, HIV, or HBV
* Presence of implantable device that is sensitive to radio frequencies ( e.g. pacemakers)
* History of autoimmune disorder, or an immunosuppressive disorder
* Stool sample with occult blood at baseline
* Any other medical, psychiatric, social condition, or occupation, in the judgement of the investigator is a contraindication to the compliance of the protocol or informed consent

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  Frequency and magnitude of adverse events

SECONDARY OUTCOMES:
Immunogenicity | 1 year
  Antibody and T cell responses to HA

CONTACTS AND LOCATIONS:
Overall Officials: Walter Doll, PhD, Principal Investigator — Scintipharma; David Liebowitz, MD, PhD, Study Director — Vaxart, Inc.
Locations (1):
- Scintipharma, Lexington, Kentucky, United States